CLINICAL TRIAL: NCT01489228
Title: Phase 2 Randomized, Multicenter, Placebo-controlled, Safety and Efficacy Study to Evaluate Three Oral E1224 Dosing Regimens and Benznidazole for the Treatment of Adult Patients With Chronic Indeterminate Chagas Disease
Brief Title: Proof-of-Concept Study of E1224 to Treat Adult Patients With Chagas Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-CH-E1224-001
Record Dates: First submitted 2011-11-24; First posted 2011-12-09 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Chagas Disease, Indeterminate
Keywords: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — Prodrugs; benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- High Dose E1224 (Experimental): High Dose (HD - 8weeks) Group
  Interventions: Drug: E1224
- Low Dose E1224 (Experimental): Low Dose (LD - 8 weeks) Group
  Interventions: Drug: E1224
- Short Dose E1224 (Experimental): Short Dose (SD - 4 weeks) Group
  Interventions: Drug: E1224
- Placebo (Placebo Comparator): Placebo (8 weeks) Group
  Interventions: Drug: Placebo
- Benznidazol (Active Comparator): BZN (Laboratório do Estado de Pernambuco -LAFEPE, tablet 100mg), 5 mg/Kg/day PO divided in two daily doses, for 60 days
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: E1224 — 100 mg tablets
  Other Names: E1224 (prodrug for active ingredient Ravuconazole)
  Arms: High Dose E1224; Low Dose E1224; Short Dose E1224
Drug: Benznidazole — 100mg tablets
  Other Names: Benznidazole (N-benzil-2-nitro-1-imidazolacetamida)
  Arms: Benznidazol
Drug: Placebo — tablets
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of E1224, a pro-drug of ravuconazole, in individuals with chronic indeterminate Chagas disease recruited in research centres in Tarija and Cochabamba, Bolivia.

DETAILED DESCRIPTION:
Chagas disease (CD) ranks among the world's most neglected diseases. In Latin America, 21 countries are endemic for CD with an estimated 108 million people at risk of contracting the disease. Estimates from the 1980s indicated that some 16 million to 18 million individuals were infected. In the 1990s, after a series of multinational control initiatives, estimates of the number of infected people were revised to 9.8 million in 2001. The estimated burden of disease in terms of disability-adjusted life years (DALYs) declined from 2.7 million in 1990 to 586,000 in 2001. Recent estimates from Pan American Health Organization (PAHO, 2006) indicate 7.54 million infected people and 55,185 new cases per year.

The only two medicines available - benznidazole (BZN) and nifurtimox (NFX) - are known to cause serious toxicity with unsatisfactory cure rates, especially when used in adult chronic CD patients.

Novel antifungal triazole derivatives have arisen as alternative treatments for CD. They inhibit T. cruzi ergosterol biosynthesis, which is essential for parasite growth and survival, and have pharmacokinetic properties suitable for the treatment of this disseminated intracellular infection. Several triazole derivatives have been tested in animal models of CD, including D08701, posaconazole, ravuconazole (RAV), albaconazole, and TAK-187. In particular, RAV has previously been shown to have potent in vitro and in vivo activities, inducing parasitological cure in mice with acute infections, including those caused by benznidazole-resistant strains of T. cruzi. Suppressive activity was also seen in dog models.

E1224 is a water-soluble monolysine salt form of the RAV pro-drug. It is a broad-spectrum triazole antifungal with in vitro activity against most Candida and Aspergillus species, some non-Aspergillus species of filamentous fungi, Cryptococcus, dermatophytes, and fungi that cause the endemic mycoses.

RAV was evaluated extensively in animal models and in human trials including Phase 2 safety and efficacy trials in oropharyngeal and esophageal candidiasis and onychomycosis, and for prevention of invasive fungal infections in hematopoietic stem cell transplant recipients.

With the benign safety profile and the encouraging results of animal studies and favorable pharmacokinetics, E1224 is considered a priority candidate for clinical development for the treatment of Chagas' disease.

The general objective of this phase II trial is to determine whether each of three different dosing regimens of E1224 are efficacious and safe in eradicating T. cruzi parasitemia in individuals with the chronic indeterminate form of CD, in comparison to placebo.

ELIGIBILITY:
Screening Criteria:

* Age >18 to < 50 years
* Weight > 40 kg
* Diagnosis of T. cruzi infection by conventional serology (a minimum of two out of three positive tests [enzyme linked immunosorbent assay (ELISA), indirect immunofluorescence (IIF), or hemagglutination inhibition (HAI)])
* Signed, written informed consent form
* No signs and/or symptoms of the chronic cardiac and/or digestive form of CD
* No acute or chronic health conditions that may interfere with the efficacy and/or safety evaluation of the study drug
* No formal contraindication to BZN and E1224
* No known history of hypersensitivity, allergic, or serious adverse reactions to the study drugs
* No history of CD treatment with BZN or NFX at any time in the past
* No history of systemic treatment with itraconazole, ketoconazole, posaconazole, isavuconazole, or allopurinol in the past

Inclusion Criteria:

* Confirmed diagnosis of T. cruzi infection by serial qualitative PCR AND Conventional serology
* Women in reproductive age must have a negative serum pregnancy test at screening, must not be breastfeeding, and consistently use and/or have partner consistently use an adequate contraceptive method
* Normal ECG at screening

Exclusion Criteria:

* Abnormal laboratory test values at screening for the following parameters: total White Blood Cells (WBC) count, platelet count, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, or creatinine; or gamma-glutamyl transferase (GGT)
* History of alcohol abuse or any other drug addiction (as specified in the Study Manual of Operations)
* Any condition that prevents the patient from taking oral medication
* Any concomitant use of antimicrobial or antiparasitic agents

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Serial negative qualitative Polymerase Chain Reaction (PCR) results (3 negative PCR results from 3 samples to be collected over 7 days) as a measure of parasitological cure at end of treatment | Day 65 (end of treatment)
  To determine whether at least one of three dosing regimens of orally administered E1224 is more efficacious than placebo in individuals with chronic indeterminate CD, by determining the number of patients who convert from positive to negative in serial, qualitative PCR test results

SECONDARY OUTCOMES:
Consistently negative serial qualitative PCR as a measure of sustained parasitological eradication | 4, 6 and 12 months follow-up
Qualitative PCR as a measure of parasite eradication | Day 8, 15, 36 , 65 and at 4, 6 and 12 months follow-up
Quantitative PCR as a measure of change in parasite load over time | Day 8, 15, 36, 65 and at 4, 6 and 12 months follow-up
Incidence of serological conversion to negative and changes in titers over time as measured by conventional and non-conventional serologies | Day 65 and at 4, 6 and 12 months after treatment
Changes in the levels of biomarkers over time: brain natriuretic peptide, troponin T, selected prothrombotic factors, lytic antibodies, apolipoprotein A1 and multiplex serodiagnostic assay | Day 36 , 65 and at 4, 6 and 12 months follow-up
Area under the plasma concentration versus time curve (AUC), Peak Plasma Concentration (Cmax), Minimum Plasma Concentration (Cmin), Clearance, Volume of Distribution , and Plasma Terminal Half-Life (t1/2) of ravuconazole and benznidazole | Day 0 (pre-dose), Day 1 (after 1st dose), Day 2, Day 3, steady-state phase (D8-D50), at the end of treatment (D65) and at the 4 months follow-up visit
  Samples for population pharmacokinetics parameters of ravuconazole and benznidazole will be collected at randomly selected time points on Days 1, 2 and 3.
Incidence and severity of adverse events (clinical and laboratory) | Up to 12 months follow-up
Incidence of Serious Adverse Events and/or adverse events leading to treatment discontinuation | Up to 12 months follow-up
Early and late predictors of sustainable response to treatments | Up to 12 months follow-up
Correlation of pharmacokinetic parameters with parasitological response, changes in biomarkers and safety outcomes | Day 8, 15, 36, 65, and at 4, 6 months and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Isabela Ribeiro, MD, Study Director — Drugs for Neglected Diseases initiative; Faustino Torrico, PhD, Principal Investigator — Universidad Mayor San Simón. Cochabamba, Bolivia.; Joaquim Gascón, PhD, Principal Investigator — CRESIB - Centre de Recerca en Salut Internacional de Barcelona, Spain.
Locations (2):
- Bolivia (2):
  - Plataforma de Atención Integral a los Pacientes con Enfermidad de Chagas, Cochabamba, Departamento de Cochabamba
  - Plataforma de Atención Integral a los Pacientes con Enfermidad de Chagas, Tarija, Tarija Department

REFERENCES:
- [Derived] De Salazar PM, Sosa-Estani S, Salvador F, Sulleiro E, Sanchez-Montalva A, Ribeiro I, Molina I, Buckee CO. Human Trypanosoma cruzi chronic infection leads to individual level steady-state parasitemia: Implications for drug-trial optimization in Chagas disease. PLoS Negl Trop Dis. 2022 Nov 21;16(11):e0010828. doi: 10.1371/journal.pntd.0010828. eCollection 2022 Nov. PMID 36409773
- [Derived] Parrado R, Ramirez JC, de la Barra A, Alonso-Vega C, Juiz N, Ortiz L, Illanes D, Torrico F, Gascon J, Alves F, Flevaud L, Garcia L, Schijman AG, Ribeiro I. Usefulness of Serial Blood Sampling and PCR Replicates for Treatment Monitoring of Patients with Chronic Chagas Disease. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01191-18. doi: 10.1128/AAC.01191-18. Print 2019 Feb. PMID 30509941
- [Derived] Torrico F, Gascon J, Ortiz L, Alonso-Vega C, Pinazo MJ, Schijman A, Almeida IC, Alves F, Strub-Wourgaft N, Ribeiro I; E1224 Study Group. Treatment of adult chronic indeterminate Chagas disease with benznidazole and three E1224 dosing regimens: a proof-of-concept, randomised, placebo-controlled trial. Lancet Infect Dis. 2018 Apr;18(4):419-430. doi: 10.1016/S1473-3099(17)30538-8. Epub 2018 Jan 16. PMID 29352704
- See also: Drugs for Neglected Diseases initiative — http://www.dndi.org